CLINICAL TRIAL: NCT06022770
Title: Clinical Study on Nutrition Intervention to Improve Nutrition and Quality of Life in Patients With Esophageal and Gastric Cancer Treated With Chemotherapy
Brief Title: Clinical Study on Nutrition Intervention in Patients With Esophageal and Gastric Cancer Treated With Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HunanCH-50
Record Dates: First submitted 2023-07-11; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Nutrition Aspect of Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Counseling (No Intervention)
- Nutrition Support Therapy (Experimental)
  Interventions: Dietary Supplement: Nutritional counseling，Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Nutritional counseling，Enteral Nutrition — patients with esophageal cancer and gastric cancer undergoing chemotherapy were selected as the study objects for nutritional risk screening, malnutrition assessment and quality of life assessment. Randomly enter the nutrition consultation group (NC) and nutrition support treatment group (NST)
  Arms: Nutrition Support Therapy

SUMMARY:
Patients with esophageal cancer and gastric cancer undergoing chemotherapy were selected as research objects to conduct nutritional risk screening, malnutrition assessment and quality of life assessment. They were randomized into the nutrition counseling group (NC) and the nutrition support therapy group (NST). To evaluate the nutrition and life quality of patients with esophageal cancer and gastric cancer before and after chemotherapy, and to study the effects of nutritional support therapy on nutrition and life quality.

DETAILED DESCRIPTION:
In view of the high incidence of malnutrition in esophageal cancer and gastric cancer and chemotherapy may further aggravate malnutrition and reduce quality of life. According to the inclusion criteria, 280 patients with esophageal cancer and gastric cancer undergoing chemotherapy were selected as research objects to conduct nutritional risk screening, malnutrition assessment and quality of life assessment. They were randomized into the nutrition counseling group (NC) and the nutrition support therapy group (NST). To evaluate the nutrition and life quality of patients with esophageal cancer and gastric cancer before and after chemotherapy, and to study the effects of nutritional support therapy on nutrition and life quality; On this basis, a nutrition and life quality management system for patients with tubular upper digestive tract chemotherapy tumors was constructed, and the system was objectively evaluated from the clinical point of view, so as to provide a feasible scheme for improving the nutrition and life quality of patients with tubular upper digestive tract chemotherapy tumors.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal or gastric cancer confirmed by histology or cytology;
* Age 18-75 years old, gender unlimited;
* Blood routine: hemoglobin ≥90g/L, absolute neutrophil count (ANC) ≥1.5×109/L, platelets ≥100×109/L; (2) Liver and kidney function: alanine transaminase（ALT）, glutamic-oxalacetic transaminease（AST）≤2.5 times the normal upper limit (with liver metastasis ≤5 times the normal upper limit); ALP≤2.5 times the normal upper limit (≤5 times the normal upper limit for patients with liver or bone metastasis); Serum total bilirubin (TBIL) was less than 1.5 times the normal upper limit. Serum creatinine (SCr) < 1.5 times the upper limit of normal; ③ Blood biochemistry: Serum albumin (ALB) ≥30g/L;
* Predicted survival of more than 3 months; It is planned to continue chemotherapy for >3 cycles in the hospital or outpatient department
* All patients participated in this study voluntarily and signed informed consent.

Exclusion Criteria:

* Other tumors, including pancreatic cancer, liver cancer and other solid digestive tract tumors, colon cancer, rectal cancer and other tubular lower digestive tract tumors;
* Have serious heart, lung and brain diseases; Complicated with chronic hepatitis, cirrhosis, chronic nephritis, renal insufficiency, etc.
* Fever associated with infection; Have difficult-to-control diabetes or other metabolic diseases;
* Patients with unstable vital signs and multiple organ failure;
* The patient has poor cognitive ability and is unable to answer questions or fill out questionnaires.
* The investigator believes that the subjects have a history of other serious systemic diseases or are not suitable for participating in this clinical study for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional risk screening（NRS） 2002 scale | Nutritional risk screening（NRS） 2002 scale during day 1 and day 42
  Nutritional risk screening（NRS） 2002 scale of patients with esophageal and gastric cancer before and after chemotherapy. The score includes 0,1,2,3,4,5,6 and 7.

SECONDARY OUTCOMES:
rates of malnutrition of patients | rates of malnutrition of patients during day 1 and day 42
  Rates of malnutrition of patients with esophageal and gastric cancer before and after chemotherapy. The result is shown as "percent".
quality of life of patients with esophageal and gastric cancer before and after chemotherapy | rates of quality of life of patients during day 1 and day 42
  quality of life of patients with esophageal and gastric cancer before and after chemotherapy. The scale include EQ-5D (score of 0-1）
quality of life of patients with esophageal and gastric cancer before and after chemotherapy | rates of quality of life of patients during day 1 and day 42
  quality of life of patients with esophageal and gastric cancer before and after chemotherapy. The scale include EQ-5D VAS (score of 1-100）

IPD SHARING:
Plan to Share IPD: No